CLINICAL TRIAL: NCT06036836
Title: A Multicenter, Randomized, Double-Blind, Phase 2, Basket Study of MK-4280A, a Coformulation of Favezelimab (MK-4280) With Pembrolizumab (MK-3475) in Selected Solid Tumors (KeyForm-010)
Brief Title: Study of Favezelimab Coformulated With Pembrolizumab (MK-4280A) in Participants With Selected Solid Tumors (MK-4280A-010)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4280A-010; MK-4280A-010 (Other: MSD); 2023-505022-34-00 (Registry Identifier: EU CT); U1111-1290-7288 (Registry Identifier: UTN)
Record Dates: First submitted 2023-08-21; First posted 2023-09-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor; Cutaneous Squamous Cell Carcinoma; Endometrial Cancer
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death-2 (PD2, PD-2); Programmed Cell Death Receptor Ligand 1 (PDL1, PD-L1); Programmed Cell Death Receptor Ligand 2 (PDL2, PD-L2); Lymphocyte-Activation Gene 3 (LAG-3)
MeSH Terms: conditions — Endometrial Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Favezelimab/Pembrolizumab (Experimental): Participants will receive coformulated favezelimab/pembrolizumab (800 mg/200 mg) via an intravenous (IV) infusion every 3 weeks (Q3W) for 3 cycles in the neoadjuvant period and 14 cycles of adjuvant therapy. Each cycle is 21 days. Participants who do not complete all 3 neoadjuvant cycles should have additional cycles in the adjuvant period so that the total number of study intervention administrations is 17 treatment cycles.
  Interventions: Biological: favezelimab/pembrolizumab
- Pembrolizumab (Experimental): Participants will receive 200 mg pembrolizumab via an IV infusion Q3W for 3 cycles in the neoadjuvant period and 14 cycles of adjuvant therapy. Each cycle is 21 days. Participants who do not complete all 3 neoadjuvant cycles should have additional cycles in the adjuvant period so that the total number of study intervention administrations is 17 treatment cycles.
  Interventions: Biological: pembrolizumab
- Favezelimab/Pembrolizumab + Lenvatinib (Cohort B) (Experimental): Participants will receive coformulated favezelimab/pembrolizumab (800 mg/200 mg) via IV infusion Q3W for up to 35 cycles (each cycle is 21 days) PLUS lenvatinib every day (QD) 20 mg orally until disease progression, unacceptable toxicity, or discontinuation criteria are met.
  Interventions: Biological: favezelimab/pembrolizumab; Drug: lenvatinib
- Pembrolizumab + Lenvatinib (Cohort B) (Experimental): Participants will receive 200 mg pembrolizumab via IV infusion Q3W for up to 35 cycles (each cycle is 21 days) PLUS lenvatinib QD 20 mg orally until disease progression, unacceptable toxicity, or discontinuation criteria are met.
  Interventions: Biological: pembrolizumab; Drug: lenvatinib

INTERVENTIONS:
Biological: favezelimab/pembrolizumab — IV infusion
  Other Names: MK-4280A
  Arms: Favezelimab/Pembrolizumab; Favezelimab/Pembrolizumab + Lenvatinib (Cohort B)
Biological: pembrolizumab — IV infusion
  Other Names: MK-3475; Keytruda®
  Arms: Pembrolizumab; Pembrolizumab + Lenvatinib (Cohort B)
Drug: lenvatinib — Oral administration of capsule
  Arms: Favezelimab/Pembrolizumab + Lenvatinib (Cohort B); Pembrolizumab + Lenvatinib (Cohort B)

SUMMARY:
The purpose of this study is to evaluate pathologic complete response (pCR) rate of coformulated favezelimab/pembrolizumab (MK-4280A) or pembrolizumab as assessed by blinded central pathology review (BICR) in participants with cutaneous squamous cell carcinoma (cSCC) [Cohort A] and to evaluate lenvatinib in combination with coformulated favezelimab/pembrolizumab or pembrolizumab with respect to objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by investigator in participants proficient in mismatch repair (pMMR) endometrial cancer (EC) [Cohort B].

ELIGIBILITY:
Inclusion Criteria

Cohort A only

* Histologically confirmed diagnosis of resectable cutaneous squamous cell carcinoma (cSCC) as the primary site of malignancy (metastatic skin involvement from another primary cancer or from an unknown primary cancer is not permitted)
* Stage II to Stage IV disease without distant metastasis (M1). cSCC tumors arising in the head and neck will be staged according to American Joint Committee on Cancer (AJCC) Edition (Ed.) 8 and cSCC tumors arising in non-head and neck locations will be staged according to Union for International Cancer Control (UICC) Ed. 8
* Is systemic treatment naïve
* Archival tumor tissue sample, or newly obtained surgical resection, or biopsy sample of a tumor lesion not previously irradiated has been provided
* Is an individual of any sex/gender, at least 18 years of age at the time of providing the informed consent

Cohort B only

* Histologically confirmed diagnosis of endometrial cancer (EC) that is not deficient in mismatch repair (dMMR) proficient in mismatch repair (pMMR) as documented by a local test report
* Documented evidence of stage IVB (per 2009 International Federation of Gynecology and Obstetrics (FIGO) staging), recurrent, or metastatic EC, and are not candidates for curative surgery or radiation
* Has radiographic evidence of disease progression after 1 prior systemic, platinum-based chemotherapy regimen for EC in any setting
* Measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST 1.1) by investigator (before first dose of study intervention)
* Is assigned female sex at birth, at least 18 years of age at the time of providing the informed consent
* Has adequately controlled blood pressure without antihypertensive medication

All Cohorts

* Agrees to follow contraception guidelines if a participant of childbearing potential
* Has a life expectancy >3 years per investigator assessment
* Has adequate organ function
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* If positive for hepatitis B, has received antiviral therapy for ≥4 weeks and undetectable viral load prior to randomization
* If positive for hepatitis C, has undetectable viral load at screening
* If positive for human immunodeficiency virus (HIV), has well-controlled HIV on a stable highly active antiretroviral therapy

Exclusion Criteria:

All Cohorts

* Has known hypersensitivity to active substances or their excipients including previous clinically significant hypersensitivity reaction to treatment with other monoclonal antibody (mAb)
* History of allogeneic tissue/solid organ transplant

Cohort A only

* Received prior radiotherapy to the index lesion (in-field lesion)
* Participants for whom the primary site of cSCC was anogenital area (penis, scrotum, vulva, perianal region) are not eligible

Cohort B

* Has had major surgery within 3 weeks prior to first dose of study interventions
* Has preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula
* Has urine protein ≥1 g/24 hours
* Has a left ventricle ejection fraction (LVEF) below the institutional (or local laboratory) normal range, as determined by multi-gated acquisition (MUGA) or echocardiogram (ECHO)
* Has radiographic evidence of encasement or invasion of a major blood vessel, or of intratumoral cavitation
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cohort A Only - Participant is an individual of any sex/gender
  Cohort B Only - Participant is assigned female sex at birth
Enrollment: 160 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate - Cohort A | Up to approximately 22 months
  Clinical benefit rate is defined as the percentage of participants who have clinical benefit. Clinical benefit is defined as major pathologic response (mPR) or pCR in participants who undergo surgery, or clinical complete response (cCR) [defined as residual tumor not visible on clinical exam nor on imaging and a negative biopsy, if biopsy is available, in participants who decline surgery.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by Investigator - Cohort B | Up to approximately 21 months
  The ORR is defined as the percentage of participants who have an OR per investigator assessment. The OR is defined as a Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.

SECONDARY OUTCOMES:
Pathologic Complete Response (pCR) - Cohort A | Up to approximately 22 months
  pCR is defined as complete absence of viable tumor in the surgical resection sample as assessed by local review of the pathology results. Number of Cohort A participants with pCR will be reported.
Major Pathologic Response (mPR) - Cohort A | Up to approximately 22 months
  mPR is defined as the presence of ≤10% of viable tumors in the surgical resection sample as assessed by local review of the pathology results. The number of Cohort A participants with mPR will be reported.
ORR per RECIST 1.1 as assessed by Investigator - Cohort A | Up to approximately 22 months
  The ORR is defined as the percentage of participants who have an OR per investigator assessment. The OR is defined as a Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.
Number of participants with an adverse event (AE) - Cohorts A and B | Up to approximately 41 months
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants who experience an AE will be reported.
Number of participants discontinuing from study therapy due to AE - Cohorts A and B | Up to approximately 41 months
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants who discontinue study treatment due to an AE will be reported.
Number of participants experiencing perioperative complications - Cohort A | Up to approximately 18 weeks
  The number of participants who experience perioperative complications will be assessed.
Number of participants with an AE that precludes surgery - Cohort A | Up to approximately 2 months
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of Cohort A participants with an AE that precludes surgery will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (44):
- United States (8):
  - Yale-New Haven Hospital-Yale Cancer Center ( Site 0643), New Haven, Connecticut
  - Dana-Farber Cancer Institute ( Site 0642), Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey ( Site 0635), New Brunswick, New Jersey
  - Duke Cancer Institute ( Site 0641), Durham, North Carolina
  - Cleveland Clinic Main ( Site 0639), Cleveland, Ohio
  - St. Luke's University Health Network ( Site 0636), Bethlehem, Pennsylvania
  - UPMC Hillman Cancer Center ( Site 0644), Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center-CRO-Simmons Comprehensive Cancer Center ( Site 0645), Dallas, Texas
- Australia (6):
  - St Vincent's Hospital-The Kinghorn Cancer Centre ( Site 0005), Darlinghurst, New South Wales
  - Royal North Shore Hospital ( Site 0008), St Leonards, New South Wales
  - Blacktown Hospital ( Site 0003), Sydney, New South Wales
  - Royal Brisbane and Women's Hospital ( Site 0002), Brisbane, Queensland
  - The Alfred Hospital ( Site 0004), Melbourne, Victoria
  - Fiona Stanley Hospital ( Site 0006), Murdock, Western Australia
- Canada (6):
  - Sunnybrook Research Institute ( Site 0607), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0606), Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal ( Site 0602), Montreal, Quebec
  - Jewish General Hospital ( Site 0605), Montreal, Quebec
  - McGill University Health Centre ( Site 0604), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0, Québec, Quebec
- France (4):
  - Institut de cancérologie Strasbourg Europe (ICANS) ( Site 0153), Strasbourg, Alsace
  - CENTRE LEON BERARD ( Site 0151), Lyon Cedex08, Auvergne-Rhône-Alpes
  - Centre Hospitalier Régional Universitaire de Brest - Hôpital Morvan ( Site 0154), Brest, Finistere
  - Hopitaux Universitaires Paris Centre-Hopital Cochin ( Site 0155), Paris
- Germany (3):
  - Universitaetsklinikum Essen ( Site 0185), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Essen-Klinik für Dermatologie, Venerologie und Allergologie ( Site 0182), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Klinik und Poliklinik für Dermatologie ( Site 0183), Dresden, Saxony
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori-SC Oncologia Medica 3 - Tumori Testa-collo ( Site 025, Milan, Lombardy
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-s.c. melanoma, immunoterapia oncologica e terapi, Napoli
- Malaysia (3):
  - Hospital Sultan Ismail-Pusat Rawatan Radioterapi Dan Onkologi ( Site 0063), Johor Bahru, Johor
  - University Malaya Medical Centre ( Site 0061), Lembah Pantai, Kuala Lumpur
  - Sarawak General Hospital-Radiotherapy Unit ( Site 0062), Kuching, Sarawak
- Netherlands (3):
  - Radboudumc ( Site 0274), Nijmegen, Gelderland
  - Erasmus Medisch Centrum ( Site 0272), Rotterdam, South Holland
  - University Medical Center Groningen ( Site 0273), Groningen
- Taiwan (3):
  - Taichung Veterans General Hospital-GYNECOLOGY ( Site 0033), Taichung
  - National Cheng Kung University Hospital-Clinical Trial Center ( Site 0032), Tainan
  - National Taiwan University Hospital ( Site 0031), Taipei
- Turkey (Türkiye) (6):
  - Medipol Mega Universite Hastanesi-oncology ( Site 0425), Stanbul, Istanbul
  - Gulhane Egitim Arastirma Hastanesi-Onkoloji ( Site 0424), Ankara
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 0421), Ankara
  - Liv Hospital Ankara-Oncology ( Site 0426), Ankara
  - Ankara Bilkent Şehir Hastanesi ( Site 0427), Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 0423), Istanbul

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26119&tenant=MT_MSD_9011